CLINICAL TRIAL: NCT00152555
Title: Physical Therapy for Improvement of Quality of Life in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Physical Therapy for Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study completed
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13238B
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2007-04

CONDITIONS: Lupus Erythematosus, Systemic; SLE
Keywords: SLE,; exercize,; physical therapy,; Systemic lupus erythematosus; relaxation therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Physical Therapy Modalities; Relaxation Therapy

INTERVENTIONS:
Behavioral: Physical Therapy or Relaxation Therapy

SUMMARY:
The purpose of this study is to see if there is an improvement in patient's quality of life, pain, and fatigue after undergoing a supervised exercise program. If improvement is found, this will help guide standard of care with lupus patients with a focus on exercise for improvement of endurance, pain and overall health.

DETAILED DESCRIPTION:
After patients have been selected and consented for this study, they will fill out a series of questionnaires. These surveys are used to stratify the patient's disease activity, assess perception of disease limitations including quality of life, fatigue and pain. We intend to use the Systemic Lupus Disease Activity Index (SLEDAI) to quantify disease activity and the SLICC to characterize the study population.

Pain, fatigue and depression will be assessed with the Pain Visual analogue scale, Fatigue Severity Score (FSS), Patient Global Assessment and BECK depression scale. Other initial data to be collected include patient's prednisone dose and resting heart rate. No specific laboratory data will be collected for this study. Patients will continue with standard of care monitoring based on their disease activity and medications.

The 100 patients will be randomized approximately 50 in the exercise group and 50 in the relaxation therapy group. The relaxation group will serve as the control arm of the study. The patients in the relaxation therapy group will then undergo a training session on biofeedback as well as receive further materials on relaxation techniques and a relaxation tape. The relaxation tape will request subjects to systematically contract and relax eleven isolated muscle groups. These muscle groups include; hands and wrists, biceps and triceps, shoulders alone, neck, tongue and mouth, eyes, nose and forehead, back alone, abdominal area alone, thighs alone, calves and feet and finally toes alone. This group of subjects will be asked to perform relaxation exercises at home a minimum of three times a week.

The subjects in the exercise group will have visits about 2 times per week for a total of 8 weeks, for a total of 16 visits. The first visit will include a general evaluation (strength, range of motion, standing balance, gait assessment, baseline vitals), determination of heart rate range for exercise and explanation of exercise portion of the study and home exercise program. Visits 2 through 16 you will participate in simple, supervised exercise at the physical therapy center at the University of Chicago. Heart rates will be measured several times throughout your exercise visits. Additionally, subjects will be asked to rate your level of pain, your blood pressure will be taken before and after and you will be advised regarding at home exercises.

Each subject will be seen for 16 visits total, unless a he/she stops attending PT sessions on their own.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of SLE by ACR criteria; Age 16+ -

Exclusion Criteria:

patients with an active lupus flare, or patients with physical limitations impairing their ability to participate in physical therapy. Other groups that will be excluded are those with limiting pulmonary disease and coronary artery disease. Patients with mechanical or structural abnormalities that would prohibit exercise (i.e. avascular necrosis of a weight-bearing joint) will also be excluded. Finally, patients already participating in a regular exercise program (>1 day per week), or those with other conditions (based on the physicians discretion) which prohibit participating in physical therapy will not qualify for this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2003-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to assess quality of life with the SF-36 Physical Function Domain.

SECONDARY OUTCOMES:
Pain, fatigue and depression assessed with the Pain Visual analogue scale, Fatigue Severity Score (FSS), Patient Global Assessment and BECK depression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Utset, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States